CLINICAL TRIAL: NCT04372251
Title: Osteosynthesis of Intraarticular Calcaneal Fractures: Arthroscopically Assisted Percutaneous Technique Versus Sinus Tarsi Approach - A Randomized Controlled Multicenter Trial
Brief Title: Osteosynthesis of Intraarticular Calcaneal Fractures: Arthroscopically Assisted Percutaneous Technique Versus Sinus Tarsi Approach
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ostfold Hospital Trust (Other)
Collaborators: Oslo University Hospital (Other); Haukeland University Hospital (Other); Vestre Viken Hospital Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20/00912
Record Dates: First submitted 2020-04-29; First posted 2020-05-04 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Calcaneus Fracture
Keywords: Calcaneal fracture; Subtalar arthroscopy; Trauma; Calcaneus
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: Two-arm parallel assignment. Patients er randomized to operative treatment with either the sinus tarsi approach or percutaneous and arthroscopically assisted osteosynthesis.
Who Masked: Investigator
Masking Description: The investigators that will conduct the follow-up examinations 2 and 5 years after surgery will be blinded for the operative treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sinus tarsi approach (STA) (Active Comparator): Patients randomized to this arm are operated with plate osteosynthesis via the sinus tarsi approach
  Interventions: Procedure: Sinus tarsi approach (STA)
- Percutaneous Arthroscopically Assisted Osteosynthesis (PACO) (Active Comparator): Patients randomized to this arm are operated with percutaneous reduction of the fracture and osteosynthesis with screws, assisted by subtalar arthroscopy
  Interventions: Procedure: Percutaneous Arthroscopically Assisted Osteosynthesis (PACO)

INTERVENTIONS:
Procedure: Sinus tarsi approach (STA) — Osteosynthesis
  Arms: Sinus tarsi approach (STA)
Procedure: Percutaneous Arthroscopically Assisted Osteosynthesis (PACO) — Osteosynthesis
  Arms: Percutaneous Arthroscopically Assisted Osteosynthesis (PACO)

SUMMARY:
In this randomized controlled trial, the outcomes of two surgical techniques for intraarticular calcaneal fractures will be evaluated and compared.

DETAILED DESCRIPTION:
Operative treatment of calcaneal features through an extensile lateral approach (ELA) has been the gold standard over many years despite high rates of infection and soft tissue complications.

Lately, there has been a trend towards less invasive fixation methods. Minimally invasive plate osteosynthesis using the sinus tarsi approach (STA) has gained popularity during the last decade.

Furthermore, percutaneous reduction and fixation techniques have been described and used for a few decades. In the early 2000s, Rammelt et al. were the first who introduced a percutaneous technique assisted by hindfoot arthroscopy. The percutaneous and arthroscopically assisted calcaneal osteosynthesis (PACO) is applicable in Sanders II and III fractures and has been shown to provide good clinical outcomes as well as a low rate of complications.

The study is designed as a superiority study. Our hypothesis is that the percutaneous and arthroscopically assisted technique provides superior outcomes compared to the sinus tarsi approach in Sanders II and III calcaneal fractures.

ELIGIBILITY:
Inclusion Criteria:

* Dislocated intraarticular calcaneal fracture, type Sanders II or Sanders III with an intraarticular step > 2mm
* Patients between 18 and 70 years of age
* Acute presentation at one of our departments, enabling surgery within 10 days after injury

Exclusion Criteria:

* Intraarticular step of < 2mm
* Sanders IV fractures
* Open fractures
* Bilateral injuries
* Concomitant major injuries of the foot, ankle or leg that affect the rehabilitation process
* Multitraumized patients
* Previous injury or surgery of the hindfoot
* Charcot foot
* Serious medical condition that contradicts surgery
* Noncompliant patients
* Insufficient Norwegian or English language skills
* Patients not available for follow-up
* Inability to conduct the rehabilitation protocol

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2020-05-05 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2031-12 (Estimated)

PRIMARY OUTCOMES:
Manchester-Oxford Foot Questionnaire (MOxFQ) | 5 years
  Foot-Ankle specific PROM (0-100 with 0 representing the best possible outcome)

SECONDARY OUTCOMES:
American Orthopaedic Foot and Ankle Society (AOFAS) Ankle-Hindfoot score | 5 years
  Widely used foot/ankle score (0-100 with 100 representing the best possible outcome)
Calcaneus Fracture Scoring System (CFSS) | 5 years
  Calcaneal fracture specific scoring system (0-100 with 100 representing the best possible outcome)
Self-reported foot and ankle score (SEFAS) | 5 years
  Foot-Ankle specific PROM (0-48 with 48 representing the best possible outcome)
Visual Analogue Scale (VAS) for pain | 5 years
  Scores pain at rest and on activity (0-10 with 0 representing no pain)
Incidence of complications | 5 years
  Yes/no for deep or superficial infection, nerve or tendon injury, deep venous thrombosis, hardware complaints and secondary surgery
Böhler angle | 5 years
  Böhler angle pre- and post surgery as well as at follow up
Subtalar osteoarthritis | 5 years
  The presence of subtalar osteoarthritis is graded based CT scans taken at the 2 year and 5 year follow-up using the Kellgren & Lawrence classification system.
EQ-5D-5L | 5 years
  Measure of health-related quality of life. This will be evaluated at the 2-year and 5 -year follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Are Stødle, MD, Principal Investigator — Oslo University Hospital; Frede Frihagen, MD, PhD, Principal Investigator — Ostfold Hospital Trust
Locations (5):
- Norway (5):
  - Haukeland University Hospital, Bergen
  - Vestre Viken Hospital Trust - Drammen hospital, Drammen
  - Oslo university hospial, Oslo
  - Vestre Viken Hospital Trust - Bærum hospital, Sandvika
  - Østfold Hospital Trust, Sarpsborg, Østfold fylke

IPD SHARING:
Plan to Share IPD: No